CLINICAL TRIAL: NCT02058043
Title: Study of MRI 3 Tesla Using Arterial Spin Labeling (Without Infusion) in Cognitive Atypical Disorders and Comparison to FDG-PET
Brief Title: Study of MRI 3Tesla Infusion Without Arterial Spin Labeling Injection (ASL) in Cognitive Atypical and Comparison to the FDG-PET
Acronym: ASLDEM DS
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-A00147; LOC1202 Gauvrit ASLDEM DS (Other: Rennes University Hospital)
Record Dates: First submitted 2013-04-05; First posted 2014-02-07 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Atypical Cognitive Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
DESCRIPTION OF RELATED QUESTION Cognitive disorders are frequently encountered and present a major public health problem given the aging of the population.

There is not one, but several neurodegenerative pathologies individual differentiated.

Particularly distinguished is Alzheimer's disease (the most common), dementia lobar fronto-temporal associated with semantic dementia (a disease with a particular tropism for semantic memory and the anterior temporal lobe), and dementia with Lewy bodies.

To differentiate these pathologies is, for the clinician, is a major issue and the clinic may not be enough.

The management and current diagnostics of atypical cognitive disorders, that is to say, patients with clinical symptoms or neuropsychological testing results suggestive of a neurodegenerative disorder other than Alzheimer's disease, are based largely on data imaging.

In the first intention, conducting imaging by MRI is recommended by the HAS, particularly to search for treatable causes to these cognitive disorders (tumors, intracranial hemorrhage in particular) but also to study the distribution of cerebral atrophy.

The sequences used are the sequences 3D T1, axial Flair, gradient echo axial T2 and coronal T2 in the plane of hippocampi and also diffusion imaging.

Research has shown interest in the study of cerebral perfusion in cognitive disorders.

The HAS recommends not to inject contrast medium on MRI in this context. The sequence of perfusion by tagging arterial protons or "arterial spin labeling" (ASL) does not use exogenous contrast medium. This is available as a commercial product, CE marked, on most of the recent clinical MRI scanners. This non-invasive technique, requiring no special precautions (e.g. verification of renal function) is used in routine clinical practice at the University Hospital of Rennes and in many centers. In the imaging of patients with dementia, it is widely used as well as the 3D T1 sequences or diffusion imaging (International Initiative ADNI) and is subject to optimization and harmonization of use in routine clinical practice with the European COST AID actions.

The second intention, an isotope imaging by FDG-PET or study of perfusion SPECT can also be performed. The interest of isotopic imaging (FDG-PET and SPECT) lies in the provision of information metabolic nonexistent in MRI, with a superiority of FDG-PET compared with SPECT. FDG-PET is the preferred examination and is carried out at CRLCC Eugène Marquis de Rennes in this context.

The aim of our study is to compare the imaging of TEPFDG, a technique not morphological, and ASL that, even if they do not study the same mode (metabolism for the first and perfusion for the second) may depict consistent anomalies.

ELIGIBILITY:
Inclusion Criteria:

* Male and females over 18 years of age
* Patients presenting with atypical cognitive disorders, clinically and through neuropsychological tests, justifying the prescription by a specialist doctor of a brain MRI and FDG-PET and lie within the context of the recommendations of the HAS.
* Patients who have received the protocol information and who given their written informed consent.

Exclusion Criteria:

Contra-indications of MRI

* Pacemaker or implantable defibrillator,
* Neurosurgical clips,
* Cochlear implants,
* Intra orbital or encephalic metallic foreign bodies,
* Endoprostheses less than 4 weeks old and osteosynthesis material used within the last 6 weeks,
* Claustrophobia. Contra-indication of FDG-PET
* Pregnancy
* Nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with atypical cognitive disorders
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
detection of hypoperfusions | less than 6 weeks
  The detection of hypoperfusions with ASL will be performed after quantification of cerebral blood flow by comparison to a template of healthy subjects of the same age.
  A base of imaging data in healthy subjects has already been acquired under another project. Some of this imaging data will be used as comparison data. No healthy subject will be included in the study ASLDEM-DS.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, IV, France